CLINICAL TRIAL: NCT06463834
Title: A Study of Sintilimab Combined With Chemotherapy for Neoadjuvant Treatment of Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FujianCH1
Record Dates: First submitted 2024-03-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Sintilimab — Sintilimab: 200mg, iv, D1, Q3W;
  DCF chemotherapy:
  docetaxel 70mg/m2，iv，d1，Q3W； cisplatin 75mg/m2，iv，d1，Q3W； 5-fluorouracil 750-800mg/m2，iv，d1-d5，Q3W
  Other Names: DCF Chemotherapy

SUMMARY:
This study is aimed to evaluate the efficacy and safety of sintilimab combined with chemotherapy (docetaxel+cisplatin+5-fluorouracil, DCF) in neoadjuvant treatment of locally advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This study was designed as a single arm, phase II trial. Subjects will receive 3 cycles of Sintilimab combined with DCF as neoadjuvant therapy. The primary endpoint is pathologic complete response(pCR).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old and ≤75 years old
* Esophageal squamous cell carcinoma diagnosed biopsy histopathology
* The primary tumor is located in the middle of the esophagus and T1b-3N1-3M0 /M1 or T3N0M0 diagnosed by CT/MRI/EUS (AJCC 8th)
* At least one measurable lesion
* Eastern cooperative oncology group (ECOG) performance status of 0 to 1
* With adequate organs function

Exclusion Criteria:

* Patients with active malignancy within 5 years other than the tumor studied in this study or a localized tumor that has been cured such as resected basal or squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, or breast cancer
* Patients who have a higher risk of bleeding or perforation due to the tumor's obvious invasion of the adjacent organs (aorta or trachea) of the esophageal lesion, or patients who have formed a fistula
* Patients who have received any anti-tumor therapy for the research disease in the past, including radiotherapy, chemotherapy, immunotherapy (including but not limited to interleukin, interferon, thymus hormone) and traditional Chinese medicine therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-03-19 (Estimated); Study Completion 2028-03-19 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 4 weeks after surgery
  Total tumor regression rate under pathologyPrimary tumor or lymph node surgery specimen pathological examination without residual tumor cell

SECONDARY OUTCOMES:
Major pathological response | 4 weeks after surgery
  Total/moderate tumor regression rate under pathologyPrimary tumor or lymph node surgery specimen pathological examination without residual tumor cell
Disease-free survival period | 3-year
  After surgery, there is no time for the disease to recur.
Incidence rate of adverse events | 3-year
  The ratio of the number of cases with adverse events to the total number of cases available for evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China